CLINICAL TRIAL: NCT02582125
Title: ONO-4538 Multicenter, Open-label, Single-arm, Phase II Study in Advanced Non-small Cell Lung Cancer
Brief Title: ONO-4538 Study in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-25
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2025-03-24 (Actual); Status verified 2024-05

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: ONO-4538; Advanced non-small cell lung cancer
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ONO-4538 (Experimental): ONO-4538 water-soluble injection, 100 mg/vial, 3 times once every 2 weeks in each 6-week cycle
  Interventions: Drug: ONO-4538

INTERVENTIONS:
Drug: ONO-4538

SUMMARY:
The objective of the study is to investigate the safety and efficacy of ONO-4538 in subjects with stage IIIB/IV or recurrent non-small cell lung cancer unsuited to radical radiotherapy and resistant to a platinum-based chemotherapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 20 years of age
* Histologically or cytologically confirmed non-small cell lung cancer
* Diagnosis of NSCLC in stage IIIB/IV unsuited to radical radiotherapy according to UICC-TNM classification (7th edition) or recurrent NSCLC
* Has at least one measurable lesion, as defined by the RECIST guideline (version 1.1)

Exclusion Criteria:

* Current or prior severe hypersensitivity to another antibody product
* Multiple primary cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse events, Laboratory tests, Vital signs, ECG, Chest X-ray, ECOG) | Approximately 6 months

SECONDARY OUTCOMES:
Response rate (centrally assessed) | Approximately 6 months
Response rate (study site assessment by investigator) | Approximately 6 months
Overall survival | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharmaceutical Co., Ltd., Study Director — Ono Pharmaceutical Co. Ltd
Locations (8):
- Taiwan (8):
  - Taichung Clinical Site 1, Taichung
  - Taichung Clinical Site 2, Taichung
  - Tainan Clinical Site 1, Tainan
  - Tainan Clinical Site 2, Tainan
  - Tainan Clinical Site 3, Tainan
  - Taipei Clinical Site 1, Taipei
  - Taipei Clinical Site 2, Taipei
  - Taipei Clinical Site 3, Taipei

REFERENCES:
- [Derived] Chen YM, Chih-Hsin Yang J, Su WC, Chong IW, Hsia TC, Lin MC, Chang GC, Chiu CH, Ho CC, Wu SY, Hung JY, Wang CC, Yang TY, Yu CJ. Nivolumab safety and efficacy in advanced, platinum-resistant, non-small cell lung cancer, radical radiotherapy-ineligible patients: A phase II study in Taiwan. J Formos Med Assoc. 2020 Dec;119(12):1817-1826. doi: 10.1016/j.jfma.2020.01.004. Epub 2020 Feb 22. PMID 32094063